CLINICAL TRIAL: NCT07168252
Title: Developing a Physiology-Pharmacodynamic Model of Rocuronium Dose and Cardiac Output to Investigate the Onset Time of Neuromuscular Relaxation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Clare Hayes-Bradley (Other)
Responsible Party: Sponsor-Investigator, Clare Hayes-Bradley, Staff Specialist Anaesthetics, Monash University
Organization: Monash University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025/PID00382 - 2025/ETH00325
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Induction of Anaesthesia; Muscle Relaxants; Rocuronium
Keywords: rocuronium; muscle relaxants; intubation
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0.6 mg/kg rocuronium IV bolus (Active Comparator)
  Interventions: Drug: Rocuronium dosing
- 1.2 mg/kg rocuronium (Active Comparator)
  Interventions: Drug: Rocuronium dosing
- 1.6mg/kg rocuronium (Experimental)
  Interventions: Drug: Rocuronium dosing
- 2.0 mg/kg (Experimental)
  Interventions: Drug: Rocuronium dosing

INTERVENTIONS:
Drug: Rocuronium dosing — Rocuronium doses of 0.6ng/kg, 1.2mg/kg, 1.6mg/kg and 2.0 mg/kg will be compared for onset speed of muscle relaxation and information on speed, cardiac output and patient body size entered into a computer model

SUMMARY:
After a patient is put to sleep, a breathing tube is often placed through the larynx (voice box) into the trachea (windpipe). To place a breathing tube requires the muscles of the jaw, voice box, and diaphragm to be relaxed. This relaxation is usually done with muscle relaxant drugs and called paralysis. Which paralysis drug and what dose should be used has been the subject of many studies.

In certain situations it is important for the patient to be fully paralysed before being intubated. Trying to intubate a partially paralysed person may result in coughing that could spread aerosols (e.g. COVID-19), patient desaturation (dropping oxygen levels), greater physiological response to intubation (heart rate, blood pressure and intra-cranial pressure rises) as well as expose the patient to risk of harm through repeated intubation attempts.

Current standard practice for patients needing critical care is to use the drug rocuronium at 1-1.2 mg/kg and wait 60 seconds for paralysis to occur. Unfortunately, 1.2mg/kg rocuronium often fails to provide good intubating conditions at 60s in some patients. The early studies revealed that 1 mg/kg rocuronium paralysis at 60s to be 'adequate' rather than 'excellent', as judged by those doing the intubation. One suggestion from 2000, was that a dose of 1.8 - 2.3 mg/kg rocuronium may be required to achieve 'excellent' intubating conditions at 60s in the vast majority of patients as is necessary clinically. The question of whether larger doses might be better has not been further investigated.

One of the reasons that the paralysis does not seem to work as fast in some patients may be related to the speed with which the drug travels round the body, pumped around the circulation, to the muscles, by the heart. This speed of circulation called cardiac output can be measured in patients at the time of injection. It may be possible to create a mathematical model for onset of paralysis by combining the information cardiac output, patient size, rocuronium dose administered, and time to paralysis. Such a model has been started by earlier researchers. The model needs further data for completion.

Once available, the model may be able to explain how fast the onset of paralysis might be in certain cardiac outputs. It might also deduce whether giving larger doses might help speed up the onset of paralysis in those patients.

ELIGIBILITY:
Inclusion Criteria:

* General anaesthesia utilising an arterial line and rocuronium at an approved study site hospital (WSLHD - Blacktown & Mount Druitt hospitals)
* Expected procedure duration >1.5 hours
* no contraindications to rocuronium neuromuscular blockade
* no contraindications to propofol TCI anaesthesia

Exclusion Criteria:

* Unable to consent for themselves for procedure
* Need for hospital interpreter (not currently funded for research use)
* pregnancy or lactation
* BMI > 50
* neuromuscular condition (e.g. affecting muscle or neuromuscular junction)
* renal failure (eGFR <30)
* chronic liver failure diagnosis
* epilepsy or antiepileptics
* lithium
* Atrial Fibrillation/Aflutter (regular rhythm needed for cardiac output monitor)
* gentamicin administered before induction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Onset of paralysis | periprocedural
  Time for neuromuscular transmission monitor (NMT) to reach 95% suppression in seconds from rocuronium injection.

SECONDARY OUTCOMES:
Cardiac output at rocuronium injection | Periprocedural
  Arterial pulse wave analysis measured cardiac output

IPD SHARING:
Plan to Share IPD: Undecided